CLINICAL TRIAL: NCT03664232
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel Group, Multicenter Study Investigating the Efficacy, Safety, and Tolerability of JNJ-42165279 in Adolescent and Adult Subjects With Autism Spectrum Disorder
Brief Title: A Study to Investigate the Efficacy, Safety, and Tolerability of JNJ-42165279 in Adolescent and Adult Participants With Autism Spectrum Disorder
Acronym: Envision
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CR108275; 42165279AUT2001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2018-09-07; First posted 2018-09-10 (Actual); Results first posted 2025-04-23 (Actual); Last update posted 2025-04-23 (Actual); Status verified 2025-04

CONDITIONS: Autism Spectrum Disorder
MeSH Terms: conditions — Autism Spectrum Disorder | interventions — JNJ-42165279

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- JNJ-42165279 (Experimental): Participants will self-administer 25 milligram (mg) JNJ-42165279 tablets orally twice daily for 12 weeks.
  Interventions: Drug: JNJ-42165279
- Placebo (Placebo Comparator): Participants will self-administer matching placebo tablets orally twice daily for 12 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: JNJ-42165279 — Participants will receive 25 mg JNJ-42165279 orally twice daily for 12 weeks.
  Arms: JNJ-42165279
Drug: Placebo — Participants will receive a matching placebo orally twice daily for 12 weeks.
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy of JNJ-42165279 compared with placebo in the improvement of symptoms of Autism Spectrum Disorder (ASD) during 12 weeks of treatment using the Autism Behavior Inventory (ABI).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Autism Spectrum Disorder (ASD) according to Diagnostic and Statistical Manual of Mental Disorders - 5th Edition (DSM-5) criteria and made or confirmed using the Autism Diagnostic Observation Schedule, 2nd edition (ADOS-2) (minimum score of 8 [autism spectrum])
* Otherwise healthy for their age group or medically stable with or without medication on the basis of physical examination, medical history, vital signs, 12-lead electrocardiogram (ECG), and clinical laboratory tests
* Have a composite score on Kaufman Brief Intelligence Test, Second Edition (KBIT-2) of at least 60
* Must live with a parent or primary caregiver or, if not, during each week he/she must either (A) spend at least 3 hours a day for at least 4 days or, (B) spend the weekend with a parent or primary caregiver
* Any pharmacologic, diet, or behavioral intervention for ASD must have begun at least 1 month prior to the baseline visit and continue unchanged through the treatment period, or have ended at least 1 month prior to the baseline visit
* Must be able to swallow the study medication whole and self-administer medication if living independently or have a parent or caregiver be able to administer medication
* Must agree to abide by the birth control requirements during the study and for 3 months after the last dose

Exclusion Criteria:

* Current or recent history of clinically significant suicidal ideation within the past 6 months, or a history of suicidal behavior within the past year
* Use of a drug with moderate/strong cytochrome P450 (CYP)3A4 inhibiting or inducing properties at, or prior to, screening that is not discontinued at least within 1 month prior to Day 1
* History of drug or alcohol use disorder according to DSM-5 criteria within 6 months before screening or positive test result(s) for alcohol or drugs of abuse (except if related to current treatment)
* Currently taking or has taken within the past month recreational or medically prescribed cannabis

Ages: 13 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 78 (Actual)
Dates: Start 2018-11-07 (Actual); Primary Completion 2022-10-17 (Actual); Study Completion 2022-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (9):
- United States (9):
  - Harmonex Neuroscience Research, Dothan, Alabama
  - Southwest Autism Research and Resource Center, Phoenix, Arizona
  - NRC Research Institute, Orange, California
  - New York Presbyterian Hospital, New York, New York
  - Nathan Kline Institute, Orangeburg, New York
  - Cincinnati Children's Hospital Medical Center, Cincinnati, Ohio
  - Cutting Edge Research Group, Oklahoma City, Oklahoma
  - BioBehavioral Research of Austin PC, Austin, Texas
  - Seattle Children's Hospital, Seattle, Washington

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo QD: Participants enrolled prior to protocol amendment-5, received placebo matched to JNJ-42165279 tablets orally once daily (QD) from Day 1 to Day 85.
- Placebo BID: Participants enrolled after protocol amendment-5 received placebo matched to JNJ-42165279 tablets orally twice daily (BID) from Day 1 to Day 85.
- JNJ-42165279 25 mg QD: Participants enrolled prior to protocol amendment-5 received JNJ-42165279 25 milligrams (mg) tablets orally QD from Day 1 to Day 85.
- JNJ-42165279 25 mg BID: Participants enrolled after protocol amendment-5 received JNJ-42165279 25 mg tablets orally BID from Day 1 to Day 85.
Period: Overall Study
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Started | 7 | 31 | 8 | 32
Treated | 7 | 30 | 8 | 32
Completed | 7 | 26 | 7 | 27
Not Completed | 0 | 5 | 1 | 5
Not completed — Withdrawal by Subject | 0 | 1 | 0 | 1
Not completed — Adverse Event | 0 | 0 | 1 | 0
Not completed — Other-Non-compliance with study drug | 0 | 1 | 0 | 2
Not completed — Other-Unspecified | 0 | 3 | 0 | 1
Not completed — - Withdrawal by Parent/Guardian | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: The full analysis set included all randomized participants who received at least 1 dose of study agent at either dose and had both a baseline and at least 1 postbaseline efficacy assessment.
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID | Total
Number analyzed (Participants) | 7 | 30 | 8 | 31 | 76
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.4 (5.13) | 19.5 (4.62) | 23.5 (4.96) | 20.9 (5.98) | 20.8 (5.35)
Age, Customized [Count of Participants; unit: Participants]
  Adolescent: 13 to 17 Years | 0 | 12 | 2 | 12 | 26
  Adult: 18 to 35 Years | 7 | 18 | 6 | 19 | 50
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 8 | 1 | 8 | 18
  Male | 6 | 22 | 7 | 23 | 58
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
  Asian | 0 | 2 | 0 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 3 | 2 | 4 | 9
  White | 7 | 25 | 6 | 23 | 61
  More than one race | 0 | 0 | 0 | 2 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 7 | 30 | 8 | 31 | 76

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Day 85 in the Autism Behavior Inventory (ABI) Core Domain Score (Social Communication and Restrictive Behaviour)
Description: ABI:62-item questionnaire to track outcomes in autism spectrum disorder (ASD). Each item was answered on 1 of 2 possible dimensions: quality (how well person carries out particular behavior; 1 to 13 items) or frequency (how often particular behavior occurs; 14 to 62 items). Each item was rated on scale of 0 (never) to 3 (very often) for frequency and 0 (without help) to 3 (not at all) for quality. Higher score=severe symptoms/more frequency. ABI core domain score was from 2 domains: social communication (23 items; 3 sub-domains) and repetitive/restrictive behavior (RRB;15 items; 4 sub-domains). Domain and sub-domain scores: calculated as average of non-missing items (ie, sum of all non-missing items divided by number of non-missing items); scores ranged from 0 to 3, higher scores=more severe symptoms of ASD. ABI core domain score=sum of social communication and RRB domain scores divided by total number of items in these 2 domains. Negative changes in ABI core domain score=improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: The full analysis set twice daily (FAS-BID) included all randomized participants who had received at least 1 dose of study agent at the BID dose and had both a baseline and at least 1 postbaseline efficacy assessment. Here, N (number of participants analyzed) signifies participants who were analyzed for this outcome measure. As per study statistical analysis plan (SAP), data for this outcome measure was planned to be collected and analyzed only on the participants who received BID dosing.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo BID | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 25 | 26
Score on a scale | -0.20 (0.400) | -0.26 (0.274)
Statistical Analysis 1: Comparison: Placebo BID vs JNJ-42165279 25 mg BID; Test type: Superiority; p = 0.284, Mixed effects model for repeatedmeasures; Least-Squares Mean Difference = -0.05, 80% CI 2-sided [-0.17 to 0.07], Standard Error of Mean 0.09

2. Primary Outcome: Change From Baseline to Day 85 in the ABI Social Communication Domain Score
Description: ABI was 62-item questionnaire completed on a web/mobile application or on paper. It tracks outcomes in ASD. Each ABI item was answered on 1 of 2 possible dimensions, quality (how well a person carries out a particular behavior; 1 to 13 items) or frequency (how often a particular behavior occurs; 14 to 62 items). Each item was rated on scale of 0 (never) to 3 (very often) for frequency and 0 (without help) to 3 (not at all) for quality. Higher score indicated severe symptoms/more frequency. The ABI social communication domain score consisted of 23 items; with 3 sub-domains. The domain and sub-domain scores were calculated as the average of the non-missing items (ie, sum of all non-missing items divided by the number of non-missing items). For both domains and its sub-domains, scores ranged from 0 to 3 with higher scores indicating more severe symptoms of ASD. Negative change in score indicates improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: The FAS-BID included all randomized participants who had received at least 1 dose of study agent at the BID dose and had both a baseline and at least 1 postbaseline efficacy assessment. Here, N (number of participants analyzed) signifies participants who were analyzed for this outcome measure. As per study SAP, data for this outcome measure was planned to be collected and analyzed only on the participants who received BID dosing.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo BID | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 25 | 26
Score on a scale | -0.22 (0.379) | -0.27 (0.332)
Statistical Analysis 1: Comparison: Placebo BID vs JNJ-42165279 25 mg BID; Test type: Superiority; p = 0.290, MMRM; Least-Squares Mean Difference = -0.05, 80% CI 2-sided [-0.18 to 0.07], Standard Error of Mean 0.1

3. Primary Outcome: Change From Baseline to Day 85 in the ABI Repetitive/Restrictive Behavior (RRB) Domain Score
Description: ABI is 62-item questionnaire completed on a web/mobile application or on paper. It tracks outcomes in ASD. Each ABI item was answered on 1 of 2 possible dimensions, quality (how well a person carries out a particular behavior; 1 to 13 items) or frequency (how often a particular behavior occurs; 14 to 62 items). Each item was rated on scale of 0 (never) to 3 (very often) for frequency and 0 (without help) to 3 (not at all) for quality. Higher score indicated severe symptoms/more frequency. The ABI RRB domain score consisted of 15 items; with 3 sub-domains. The domain and sub-domain scores were calculated as the average of the non-missing items (ie, sum of all non-missing items divided by the number of non-missing items). For both domains and its sub-domains, scores ranged from 0 to 3 with higher scores indicating more severe symptoms of ASD. Negative change in score indicates improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo BID | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 25 | 26
Score on a scale | -0.17 (0.525) | -0.23 (0.299)
Statistical Analysis 1: Comparison: Placebo BID vs JNJ-42165279 25 mg BID; Test type: Superiority; p = 0.231, MMRM; Least-Squares Mean Difference = -0.08, 80% CI 2-sided [-0.21 to 0.06], Standard Error of Mean 0.1

4. Secondary Outcome: Change From Baseline to Day 85 in the ABI Mood and Anxiety Domain Score
Description: ABI was 62-item questionnaire to track outcomes in ASD. Each ABI item was answered on 1 of 2 possible dimensions, quality (how well a person carries out a particular behavior; 1 to 13 items) or frequency (how often a particular behavior occurs; 14 to 62 items). Each item was rated on scale of 0 (never) to 3 (very often) for frequency and 0 (without help) to 3 (not at all) for quality. Higher score indicated severe symptoms/more frequency. ABI mood and anxiety domain had 9 items with 5 sub-domains. ABI mood and anxiety domain and its sub-domains, scores ranged from 0 to 3 with higher scores indicating more severe symptoms of ASD. Domain and sub-domain scores were calculated as the average of the non-missing items (ie, sum of all non-missing items divided by the number of non-missing items). Negative changes in ABI mood and anxiety domain score indicated improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: The FAS analysis set included all randomized participants who had received at least 1 dose of study agent at either dose and had both a baseline and at least 1 postbaseline efficacy assessment. Here, N (number of participants analyzed) signifies participants who were analyzed for this outcome measure.
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 6 | 25 | 7 | 26
Score on a scale | -0.30 (0.408) | -0.23 (0.622) | -0.19 (0.551) | -0.26 (0.552)

5. Secondary Outcome: Change From Baseline to Day 85 in the ABI Challenging Behavior Domain Score
Description: ABI was 62-item questionnaire to track outcomes in ASD. Each ABI item was answered on 1 of 2 possible dimensions, quality (how well a person carries out a particular behavior; 1 to 13 items) or frequency (how often a particular behavior occurs; 14 to 62 items). Each item was rated on scale of 0 (never) to 3 (very often) for frequency and 0 (without help) to 3 (not at all) for quality. Higher score indicated severe symptoms/more frequency. ABI challenging behavior domain had 7 items with 4 sub-domains. ABI challenging behavior domain and its sub-domains, scores ranged from 0 to 3 with higher scores indicating more severe symptoms of ASD. The domain and sub-domain scores were calculated as the average of the non-missing items (ie, sum of all non-missing items divided by the number of non-missing items). Negative changes in ABI challenging behavior domain score indicated improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 6 | 25 | 7 | 26
Score on a scale | -0.27 (0.329) | -0.22 (0.533) | -0.20 (0.411) | -0.20 (0.532)

6. Secondary Outcome: Change From Baseline to Day 85 in the ABI Self-Regulation Domain Score
Description: ABI was 62-item questionnaire to track outcomes in ASD. Each ABI item was answered on 1 of 2 possible dimensions, quality (how well a person carries out a particular behavior; 1 to 13 items) or frequency (how often a particular behavior occurs; 14 to 62 items). Each item was rated on scale of 0 (never) to 3 (very often) for frequency and 0 (without help) to 3 (not at all) for quality. Higher score indicated severe symptoms/more frequency. ABI self-regulation domain had 8 items with 2 sub-domains. ABI self-regulation domain and its sub-domains, scores ranged from 0 to 3 with higher scores indicating more severe symptoms of ASD. The domain and sub-domain scores were calculated as the average of the non-missing items (ie, sum of all non-missing items divided by the number of non-missing items). Negative changes in ABI self-regulation domain score indicated improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 6 | 25 | 7 | 26
Score on a scale | -0.31 (0.272) | -0.20 (0.510) | -0.11 (0.364) | -0.18 (0.380)

7. Secondary Outcome: Change From Baseline to Day 85 in the Aberrant Behavior Checklist (ABC) Subscales Scores
Description: The ABC was 58-item behavior rating scale used to measure behavior problems across 5 subscales: irritability (15 items), lethargy (social withdrawal; 16 items), stereotypic behavior (7 items), hyperactivity/ noncompliance (16 items), and inappropriate speech (4 items). Items were rated on a 4-point scale score ranging from 0 (not at all a problem) to 3 (the problem is severe in degree). The total subscale scores ranged from 0 to 45, 0 to 48, 0 to 21, 0 to 48 and 0 to 12 for irritability, lethargy (social withdrawal), stereotypic behavior, hyperactivity, and inappropriate speech respectively. The higher scores indicating more severe behavior problems. Negative change in score indicated improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 7 | 26 | 7 | 28
Score on a scale
  Irritability | -5.86 (5.398) | -3.80 (6.408) | -2.71 (6.291) | -4.18 (8.940)
  Lethargy/Social Withdrawal | -6.86 (5.014) | -3.31 (7.092) | -2.71 (4.680) | -5.14 (7.271)
  Stereotypic Behavior | -1.86 (2.340) | -1.19 (3.359) | -0.14 (1.676) | -1.68 (3.128)
  Hyperactivity/Noncompliance | -6.00 (3.916) | -4.77 (7.010) | -2.00 (6.351) | -4.07 (6.532)
  Inappropriate Speech | -1.43 (2.573) | -0.85 (1.826) | -0.43 (0.787) | -0.86 (2.138)

8. Secondary Outcome: Change From Baseline to Day 71 in the Autism Behavior Inventory-Short Form (ABI-S) Domains Scores
Description: The ABI-S was the shorter version of ABI. It consists of 24 items across 5 areas: challenging behavior (3 items), mood and anxiety (5 items), restrictive behaviors (7 items), social communication (6 items), and self-regulation (3 items). Each item was answered on 1 of 2 possible dimensions, quality (how well a person carries out a particular behavior or frequency (how often a particular behavior occurs). Each ABI-S domain score was calculated as the sum of the scores in the ABI-S domain divided by the total number of items in this domain. Each item was rated on scales of 0 (never) to 3 (very often) for frequency and 0 (without help) to 3 (not at all) for quality. The total subscale scores ranged from 0 to 9, 0 to 15, 0 to 21, 0 to 18, and 0 to 9, for challenging behavior, mood and anxiety, restrictive behaviors, social communication, and self-regulation respectively. Lower score indicated better performance. Negative change in score indicates improvement.
Time Frame: Baseline (Day 1) to Day 71
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 5 | 18 | 5 | 22
Score on a scale
  Challenging behavior | 0.07 (0.548) | -0.17 (0.618) | -0.33 (0.707) | -0.32 (0.477)
  Mood and anxiety | -0.48 (0.782) | -0.24 (0.473) | 0.32 (0.179) | -0.21 (0.624)
  Restrictive behaviors | -0.14 (0.440) | -0.12 (0.580) | 0.11 (0.275) | -0.23 (0.383)
  Social communication | -0.37 (0.431) | -0.38 (0.520) | -0.23 (0.480) | -0.31 (0.425)
  Self regulation | -0.47 (0.506) | 0.04 (0.740) | 0.13 (0.447) | -0.29 (0.637)

9. Secondary Outcome: Change From Baseline to Day 85 in the Autism Behavior Inventory-Clinician Interview (ABI-C) Domains Scores
Description: The ABI-C covers the domains of ABI and was intended for completion by the clinician following an interview with caregiver and observation or interview with the individual with ASD, as appropriate. The ABI-C was designed to capture the behaviors of a person with ASD that have occurred over the past week. There were 14 items across each of the 5 domains: challenging behavior (2 items), mood and anxiety (2 items), restrictive behaviors (5 items), social communication (3 items), and self-regulation (2 items). The clinician rates the severity of behaviors or level of impairment on a scale of 1 (no impairment) to 7 (very severe difficulties) with a higher score indicating more severe symptoms of ASD. Total subscale scores ranged from 0 to 14, 0 to 14, 0 to 35, 0 to 21 and 0 to 14, for challenging behavior, mood and anxiety, restrictive behaviors, social communication and self-regulation respectively. Lower score indicated better performance. Negative change in score indicates improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 7 | 27 | 7 | 29
Score on a scale
  Challenging behavior | -0.64 (1.107) | -0.26 (0.739) | -0.07 (1.018) | -0.40 (1.030)
  Mood and anxiety | -0.36 (0.690) | -0.44 (0.859) | -0.07 (0.450) | -0.60 (1.270)
  Restrictive behaviors | -0.29 (0.430) | -0.47 (0.686) | -0.43 (0.582) | -0.52 (0.863)
  Social communication | 0.05 (0.300) | -0.59 (0.669) | -0.05 (0.525) | -0.70 (0.993)
  Self regulation | -0.14 (0.627) | -0.41 (1.029) | -0.07 (0.189) | -0.22 (0.862)

10. Secondary Outcome: Change From Baseline to Day 85 in the Clinical Global Impression-Severity (CGI-S) Scale Score
Description: The CGI-S 7-point scale was a global assessment that measures the clinician's impression of the severity of illness of the participant. A rating scale of 1 to 7 was used, with 1="normal, not at all ill" and 7="among the most extremely ill". Higher score indicated more severe illness.
Time Frame: Baseline (Day 1) to Day 85
Population: as for outcome 2
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Placebo BID | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 26 | 28
Score on a scale | 0.0 [-2 to 1] | 0.0 [-3 to 1]

11. Secondary Outcome: Change From Baseline to Day 85 in the Repetitive Behavior Scale - Revised (RBS-R) Subscale Score
Description: The RBS-R was a 43-item report scale to indicate the occurrence of repetitive behaviors and degree to which a behavior was a problem scored on a range between 0 (behavior did not occur) to 3 (behavior occurred and was a severe problem). There are 6 subscale scores: Stereotyped Behavior (items 1 to 6), self-injurious behavior (items 7 to 14), compulsive behavior (items 15 to 22), ritualistic behavior (items 23 to 28), sameness behavior (items 29 to 39), and restricted behavior (items 40 to 43). The ranges for RBS-R subscale scores were stereotyped behavior: 0 to 18; self-injurious behavior: 0 to 24; compulsive behavior: 0 to 24; ritualistic behavior: 0 to 18; sameness behavior: 0 to 33; and restricted behavior: 0 to 12. Higher scores indicate more severe problems with repetitive behaviors and a decrease (a negative change) from baseline represents improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 7 | 27 | 7 | 29
Score on a scale
  stereotyped behavior | -1.6 (2.07) | -0.6 (2.34) | -1.0 (1.83) | -0.8 (1.89)
  self-injurious behavior | -1.4 (1.99) | 0.2 (2.15) | -0.7 (1.60) | -1.2 (2.05)
  compulsive behavior | -1.7 (4.61) | -0.4 (2.95) | -1.0 (1.53) | -0.8 (2.33)
  ritualistic behavior | -2.6 (3.21) | -0.5 (3.71) | -1.6 (2.15) | -1.1 (3.63)
  sameness behavior | -6.3 (4.89) | -2.0 (4.98) | -2.3 (3.15) | -2.9 (6.39)
  restricted behavior | -0.4 (3.05) | -0.5 (1.83) | -0.3 (2.81) | -0.7 (2.55)

12. Secondary Outcome: Change From Baseline to Day 85 in the Zarit Burden Interview (ZBI) Global Score
Description: The ZBI short version scale consists of 22 items designed to assess the psychological burden experienced by a caregiver. Items ask how the caregiver felt and their responses range from 0 to 4, where 0 = never and 4 = nearly always. The ZBI global score was the sum of all item score and ranges from 0 to 88 with higher scores indicating a higher burden. A negative change in the ZBI global score from baseline representing improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 7 | 30 | 8 | 29
Score on a scale | -2.0 (12.12) | -2.2 (10.89) | -4.3 (7.83) | -3.9 (10.20)

13. Secondary Outcome: Change From Baseline to Day 85 in the Child Adolescent Symptom Inventory - Anxiety (CASI-Anx) Scale Score
Description: The CASI assesses symptoms of the following disorders: attention deficit hyperactivity disorder, oppositional defiant disorder, conduct disorder, generalized anxiety disorder, social phobia, separation anxiety disorder, disruptive mood dysregulation disorder, major depressive episode, manic episode, dysthymic disorder, schizophrenia, autistic/Asperger's disorder, anorexia, and bulimia. CASI-Anx scale total is a 21-point anxiety subscale of the full CASI. Responses were ranged from 0 to 3, where 0 = never and 3 = very often. The CASI-Anx scale total score ranges from 0 to 63 with higher scores indicating more severe anxiety. Negative changes in Symptom Severity scores indicate improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 7 | 27 | 7 | 29
Score on a scale | -5.14 (7.647) | -4.89 (8.135) | -1.86 (2.610) | -5.19 (8.020)

14. Primary Outcome: Change From Baseline to Day 85 in the Social Responsiveness Scale 2 (SRS-2) Total T-Score
Description: SRS-2: 65-item scale measured extent of autistic social impairment and included 5 subscales: social awareness, social cognition, social communication, social motivation, and restricted interests and repetitive behavior. Each of 65 items had 4 responses: not true, sometimes true, often true, and almost always true. Scoring value for each item was 0 to 3. If a response to an item was missing, then pre-defined median value for item (0 or 1) was imputed. SRS-2 was not scored if 7 or more item responses were missed. Total raw score was sum of item response values. Each subscale was obtained by adding response values and converted total raw score to standardized T-score based on gender and rater (parent or caregiver). Total T-score was categorized: within normal limits (<=59), mild (60 to 65), moderate (66 to 75) and severe (>=76). For total score T-score, higher scores=more severe symptoms. SRS T-score had mean of 50 and standard deviation of 10. Negative changes in T-scores=improvement.
Time Frame: Baseline (Day 1) to Day 85
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: T-score
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 7 | 27 | 7 | 29
T-score | -6.4 (4.79) | -4.6 (7.91) | -4.1 (6.99) | -7.1 (7.73)

15. Secondary Outcome: Change From Baseline to Day 85 in the Caregiver Global Impression of Severity (Caregiver GI-S) Scale Score
Description: The caregiver GI-S is a single-item instrument that asks caregivers to rate their overall impression of the severity of their child's ASD symptoms. A rating scale of 1 to 7 was used, with 1= none and 7=severe illness. Higher score indicated more severe illness.
Time Frame: Baseline (Day 1) to Day 85
Population: as for outcome 2
Measure: Median (Full Range); unit: Score on a scale
Arm/Group | Placebo BID | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 26 | 28
Score on a scale | 0.0 [-3 to 2] | 0.0 [-4 to 2]

16. Secondary Outcome: Caregiver Assessment of Treatment: Question 1: Number of Participants With Overall Status (Improvement) of Autism at Day 85
Description: The caregiver assessment of treatment is a 3-item questionnaire completed at the end of the treatment period. The first question asks caregivers to rate their overall impression of improvement in their child's autism since starting the study medication, with 7 response options ranging from 1 "very much improved" to 7 "very much worse".
Time Frame: At Day 85
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 7 | 29 | 8 | 29
Participants
  Very much improved | 0 | 2 | 0 | 3
  Much improved | 2 | 3 | 0 | 2
  Improved | 3 | 7 | 5 | 10
  No change | 2 | 15 | 3 | 13
  Worse | 0 | 1 | 0 | 1
  Much worse | 0 | 1 | 0 | 0
  Very Much Worse | 0 | 0 | 0 | 0

17. Secondary Outcome: Caregiver Assessment of Treatment: Question 2: Number of Participants With Improvement in Specific Symptoms During Treatment at Day 85
Description: The caregiver assessment of treatment was a 3-item questionnaire completed at the end of the treatment period. The second question asks caregivers whether there was improvement in 9 specific symptoms (child communicated more, child's repetitive behaviors improvement, child's restricted interests, child's mood improved, child was less anxious, child better perform daily activities, child more interest social activities, child's sleep improved, child less distracted), with responses options of Yes or No.
Time Frame: At Day 85
Population: The FAS analysis set included all randomized participants who had received at least 1 dose of study agent at either dose and had both a baseline and at least 1 postbaseline efficacy assessment. Here, N (number of participants analyzed) signifies participants who were analyzed for this outcome measure and n (number analyzed): number of participants evaluable at each specified category.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 7 | 29 | 8 | 29
Participants
  Child communicated more- No | 4 | 16 | 4 | 12
  Child communicated more- Yes | 3 | 13 | 4 | 17
  Child repetitive behaviors improvement -No: number analyzed (Participants) | 6 | 29 | 8 | 29
  Child repetitive behaviors improvement -No | 3 | 24 | 6 | 19
  Child repetitive behaviors improvement -Yes: number analyzed (Participants) | 6 | 29 | 8 | 29
  Child repetitive behaviors improvement -Yes | 3 | 5 | 2 | 10
  Child Restricted Interests Improved- No: number analyzed (Participants) | 6 | 29 | 8 | 29
  Child Restricted Interests Improved- No | 3 | 24 | 6 | 16
  Child Restricted Interests Improved- Yes: number analyzed (Participants) | 6 | 29 | 8 | 29
  Child Restricted Interests Improved- Yes | 3 | 5 | 2 | 13
  Child Mood Improved- No: number analyzed (Participants) | 7 | 28 | 8 | 29
  Child Mood Improved- No | 2 | 17 | 2 | 15
  Child Mood Improved- Yes: number analyzed (Participants) | 7 | 28 | 8 | 29
  Child Mood Improved- Yes | 5 | 11 | 6 | 14
  Child Was Less Anxious- No: number analyzed (Participants) | 7 | 28 | 8 | 29
  Child Was Less Anxious- No | 5 | 18 | 2 | 18
  Child Was Less Anxious-Yes: number analyzed (Participants) | 7 | 28 | 8 | 29
  Child Was Less Anxious-Yes | 2 | 10 | 6 | 11
  Child Better Perform Daily Activities- No | 3 | 17 | 3 | 16
  Child Better Perform Daily Activities- yes | 4 | 12 | 5 | 13
  Child More Interest Social Activities- No | 3 | 17 | 4 | 17
  Child More Interest Social Activities- Yes | 4 | 12 | 4 | 12
  Child Sleep Improved -No | 5 | 21 | 6 | 18
  Child Sleep Improved -Yes | 2 | 8 | 2 | 11
  Child Less Distracted- No: number analyzed (Participants) | 6 | 29 | 8 | 29
  Child Less Distracted- No | 5 | 24 | 5 | 19
  Child Less Distracted-Yes: number analyzed (Participants) | 6 | 29 | 8 | 29
  Child Less Distracted-Yes | 1 | 5 | 3 | 10

18. Secondary Outcome: Caregiver Assessment of Treatment: Question 3: Number of Participants With Interest in Continuing Treatment at Day 85
Description: The caregiver assessment of treatment is a 3-item questionnaire completed at the end of the treatment period. The third question asked caregivers their interest in having their child continue the study medication. There were 5 response options ranging from "Not at all interested" to "Extremely interested".
Time Frame: At Day 85
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 7 | 29 | 8 | 29
Participants
  Extremely Interested | 2 | 10 | 0 | 6
  Very Interested | 1 | 3 | 2 | 5
  Moderately Interested | 1 | 7 | 1 | 6
  A Little Interested | 2 | 4 | 3 | 4
  Not At All Interested | 1 | 5 | 2 | 8

19. Secondary Outcome: Self Global Impression of Improvement (Self GI-I) Scale Score at Day 85
Description: Self-Global impression of improvement (Self GI-I) scale score at Day 85 was reported. At the end of the treatment period, the participant was asked to give his/her impression of overall improvement in ASD symptoms using a single-item instrument, the Self GI-I. The scale ranges from 1 (very much better) to 7 (very much worse), with higher scores indicating worsening of symptoms.
Time Frame: At Day 85
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo BID | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 30 | 27
Score on a scale | 3.03 (1.098) | 3.41 (0.931)

20. Secondary Outcome: Clinical Global Impression-Improvement (CGI-I) Score (Frequency Distribution) at Day 85
Description: The CGI-I was single-item instrument that measures the clinician's global impression of improvement in the participant from the initiation of treatment. The CGI-I was 7-point scale to measure improvement in illness, where 1=very much improved, 2=much improved, 3=minimally improved, 4=no change from baseline, 5=minimally worse, 6=much worse, 7=very much worse.
Time Frame: At Day 85
Population: as for outcome 17
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
Number analyzed (Participants) | 1 | 26 | 2 | 27
Participants
  Very much improved | 0 | 0 | 0 | 0
  Much improved | 0 | 3 | 0 | 7
  Minimally improved | 1 | 9 | 0 | 5
  No change | 0 | 14 | 2 | 15
  Minimally worse | 0 | 0 | 0 | 0
  Much worse | 0 | 0 | 0 | 0
  Very much worse | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: Serious adverse events (SAEs) and other adverse events (AEs): From Day 1 up to 6 days post last dose of study drug (up to 91 days); All-cause mortality: From screening (Day -26) up to 99 days
Description: SAEs and other AEs: The safety analysis set included all randomized participants who had received at least 1 dose of study drug. All-cause mortality: all randomized analysis set included all participants who were randomized in the study (that is, participants who reported a randomization date or were assigned a randomization number) regardless of whether treatment was received.
Arm/Group | Placebo QD | Placebo BID | JNJ-42165279 25 mg QD | JNJ-42165279 25 mg BID
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/31 | 0/8 | 0/32
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/30 | 0/8 | 0/32
Other Adverse Events (participants affected / at risk) | 5/7 | 7/30 | 7/8 | 3/32
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo QD (N=7) | Placebo BID (N=30) | JNJ-42165279 25 mg QD (N=8) | JNJ-42165279 25 mg BID (N=32)
Early Repolarisation Syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Motion Sickness (Ear and labyrinth disorders) | 0 | 0 | 1 | 0
Abdominal Discomfort (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Medical Device Site Rash (General disorders) | 0 | 0 | 1 | 0
Seasonal Allergy (Immune system disorders) | 1 | 0 | 1 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 1 | 0
Nasopharyngitis (Infections and infestations) | 1 | 0 | 1 | 0
Upper Respiratory Tract Infection (Infections and infestations) | 1 | 1 | 0 | 1
Ligament Sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Alanine Aminotransferase Increased (Investigations) | 0 | 2 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Increased Appetite (Metabolism and nutrition disorders) | 1 | 1 | 0 | 0
Headache (Nervous system disorders) | 2 | 2 | 0 | 1
Lethargy (Nervous system disorders) | 0 | 0 | 1 | 0
Sedation (Nervous system disorders) | 0 | 1 | 1 | 0
Oropharyngeal Pain (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Acne (Skin and subcutaneous tissue disorders) | 1 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
If an investigator wishes to publish information from the study, a copy of the manuscript must be provided to the sponsor for review at least 60 days before submission for publication or presentation. If requested by the sponsor in writing, the investigator will withhold such publication for up to an additional 60 days to allow for filing of a patent application.

DOCUMENTS (2):
  • Study Protocol (2020-09-29): https://cdn.clinicaltrials.gov/large-docs/32/NCT03664232/Prot_000.pdf
  • Statistical Analysis Plan (2022-11-22): https://cdn.clinicaltrials.gov/large-docs/32/NCT03664232/SAP_001.pdf